CLINICAL TRIAL: NCT04336631
Title: Implementation of DCP3 Strategies to Manage and Control Hypertension Among Hypertensive Patients in Pakistan: A Randomized Controlled Trial
Brief Title: DCP3 Based Multi-component Intervention for Hypertension Management and Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Services Academy, Islamabad, Pakistan (Other)
Responsible Party: Principal Investigator, Subhana Akber Khan, Principal Investigator PhD Scholar (Public Health), Health Services Academy, Islamabad, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: NCT 2224/2017
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Hypertension; Hypertensive Patients
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Medical Follow Up, Counseling & Usual Care (Other): Behavioral counseling was provided to the patients on each consecutive follow up after enrolling in this study. They were adequately followed on physical exercise, reduced salt intake, lifestyle modifications, and smoking cessation. All measurements of blood pressure and weight were maintained and recorded.
  Interventions: Behavioral: Intervention on DCP3 based strategies for Hypertension Management and Control
- Routine Medical Follow Up & Usual Care (No Intervention): Usual routine medical care was provided to the study participants only.

INTERVENTIONS:
Behavioral: Intervention on DCP3 based strategies for Hypertension Management and Control — Intervention on DCP3 based strategies for Hypertension Management and Control was developed after formative research findings and evidence built on desk review which was conducted prior to implementation of the multi-componnet strategy. It was tested and implemented in a tertiary care hospital of cardiology among hypertensive patients visiting out-patient department in Rawalpindi, Pakistan.
  Arms: Routine Medical Follow Up, Counseling & Usual Care

SUMMARY:
This study aims to enable delivery of a multi-component intervention comprising of strategies based on Disease Control Priorities 3rd edition for management of hypertension among hypertensive patients. The secondary objective is to test the feasibility, acceptability and adaptability of a multi-component intervention delivered at a tertiary level health-care facility in the cultural context of Pakistan. A formative research study was conducted before so as to develop and test the intervention in a tertiary care hospital setting. The investigators employed qualitative research methods to explore the feasibility, applicability, and acceptance of DCP3 based intervention comprising of strategies for hypertension management. Focus group discussions and in-depth interviews with selected study participants were conducted at Armed Forces Institute of Cardiology (AFIC/NIHD), Rawalpindi for which a prior written and verbal consent was obtained from all research participants. The study adhered to the ethical principles of involving human subjects in the research. All information provided by the participants was recorded and was kept strictly confidential.

ELIGIBILITY:
Inclusion Criteria:

* • Pakistani nationals both male and female of age 18 years and above will be invited to participate in the study

  * Similarly; known hypertensive patients having a systolic blood pressure of ≥140 mmHg on current treatment will be included &
  * Patients with co-morbidities will also be included such as those suffering from cardiac ailments (angina or transient ischemic attack (TIA) and diabetes

Exclusion Criteria:

* • Patients with compromised neurological or cognitive state who are unable to provide their consent will be excluded

  * Patients suffering from non-cardiovascular diseases and life-threatening illnesses such as angiographically proven coronary disease, peripheral or cerebral vascular disease, pulmonary hypertension, having history of myocardial infarction, stroke/PCI/stent or high-risk conditions will be excluded from participation
  * Patients with chronic conditions and co-morbidities requiring surgical intervention or treatment such as cardiomyopathies or congenital abnormalities &
  * Patients receiving dialysis will also be excluded from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adequate blood pressure control in the intervention arm after delivering the intervention at 03 months | 03 months
Number of participants with reduced salt intake from baseline measurements as compared to follow up measurements at 03 months | Baseline to follow up in 03 months
  This was assessed at each consecutive follow up of hypertensive patients for reduced salt intake and increased physical exercise. Hypertensive patients were also counselled for regular intake of medicines prescribed by the physician. A record for the mentioned measurements was kept and maintained from baseline to 03 months of the trial.
Number of participants with increased level of physical exercise compared from baseline measurements to follow up measurements at 03 months | 03 months
  This was assessed at each consecutive follow up of hypertensive patients for reduced salt intake and increased physical exercise. Hypertensive patients were also counselled for regular intake of medicines prescribed by the physician. A record for the mentioned measurements was kept and maintained from baseline to 03 months of the trial.
Number of participants with regular compliance to medications from baseline measurement compared with follow up measurements at 03 months | 03 months
  This was assessed at each consecutive follow up of hypertensive patients for reduced salt intake and increased physical exercise. Hypertensive patients were also counselled for regular intake of medicines prescribed by the physician. A record for the mentioned measurements was kept and maintained from baseline to 03 months of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Armed Forces Institute of Cardiology (AFIC/NIHD), Rawalpindi, <Select>, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Khan SA, Hafeez A, Zaka A, Khan SA, Ahmed A, Pervaiz F, Siddiqui AH. A Randomized Controlled Trial of Blood Pressure Reduction Based on Disease Control Priorities 3 in Pakistan to Manage and Control Hypertension. High Blood Press Cardiovasc Prev. 2023 Jul;30(4):357-366. doi: 10.1007/s40292-023-00589-y. Epub 2023 Jul 26. PMID 37493898
- See also: A Study Protocol on Hypertension — http://www.pafmj.org/index.php/PAFMJ/article/view/3932/2548

DOCUMENTS (1):
  • Study Protocol (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04336631/Prot_000.pdf